CLINICAL TRIAL: NCT03708341
Title: Exogenous Melatonin in Intensive Care Unit Chronodisruption: Randomized Controled Trial
Brief Title: Exogenous Melatonin in Intensive Care Unit Chronodisruption
Acronym: EMIC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Saint-Joseph University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LPCQM/07/17
Record Dates: First submitted 2018-09-26; First posted 2018-10-17 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Sleep Deprivation; Intensive Care Psychosis
Keywords: melatonin; Sleep Deprivation; Intensive Care Psychosis
MeSH Terms: conditions — Sleep Deprivation | interventions — Melatonin

STUDY DESIGN:
Intervention Model Description: Randomized Controled Trial. GLMM will be used to analyze the data due to its ability to handle non-normal distributions and account for both fixed and random effects.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo, double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Melatonin (Experimental): Patients will be administered melatonin 5 mg at a fixed time every day during their ICU stay (from day of admission till day of discharge from ICU)
  Interventions: Drug: Melatonin 5 mg
- Placebo (Placebo Comparator): Patients will be administered a placebo pill that is identical in shape and color to the melatonin pill, at a fixed time every day during their ICU stay
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Melatonin 5 mg — Systematic daily administration of melatonin 5 mg during patient's ICU stay
  Arms: Melatonin
Drug: Placebo Oral Tablet — Systematic daily administration of placebo during patient's ICU stay
  Arms: Placebo

SUMMARY:
To this day, a small number of studies have evaluated the effect of melatonin on the modifications of the characteristics of sleep in critical care units, with mostly a small studied population. However, no study has been realized on a large population, nor has it evaluated the association between genetic factors and response to treatment (melatonin), hence the originality of our study. In our study we hypothesized that systematic melatonin usage in ICU can ameliorate the total sleep time and the fragmentation index and can decrease the confusion related to sleep deprivation.

DETAILED DESCRIPTION:
1. Rationale:

   1.1. Sleep and the circadian rhythm: Sleep is usually considered to be a time of rest and recovery from the stress of daily life. It also plays a crucial role in the normal immune and endocrine systems. Studies showed that there is a link between sleep duration and a large variety of health issues, including obesity, diabetes mellitus, hypertension and depression. Furthermore, sleep deprivation has been linked to immunosuppression as well as alterations in normal wound healing, thermoregulation and upper airway muscles (leading to a blunted response to hypercapnia and hypoxia).

   Sleep is divided into 2 cycles: non-REM (NREM) sleep and REM sleep. NREM sleep is divided into 4 more stages (1, 2, 3 and 4). REM sleep is characterized by the presence of rapid ocular movements, and is commonly known as the phase during which dreams occur. Most individuals progress through the various stages, starting from NREM stage 1, to finally reach REM sleep. Usually, each sleep cycle lasts 90 minutes , with an average of 4-5 cycles per night.

   During sleep, various hormonal changes occur, which shows the importance of sleep in the normal functioning of the body. Growth hormone and cortisol are released during sleep, and melatonin levels markedly increased at sleep initiation, with a decrease right before waking up. Circadian rhythms are normal fluctuations of the biological function, and are part of an endogenous 24 hour clock situation in the supra-chiasmatic nucleus (SCN) of the anterior hypothalamus, responsible for controlling the day/night variations of physiological and behavioral functions of the organism. These wake/sleep cycles are usually divided into an average of 8 hours of nocturnal sleep and 16 hours of wakefulness in humans.

   Circadian rhythms make cyclic environmental changes easier to adapt to, and influence a number of behaviors and physiological parameters. This is due to a genetic molecular clock which is present in most nucleated cells. This clock is composed of a group of transcription factors and regulators of transcription factors which exerce a retro-control over one another. Thus, protein of the molecular clock can have very important effects on the transcriptional activity and the metabolism, leading, directly or indirectly, to a variation of 50% of the total gene pool.

   1.2. Sleep disorders Sleep disorders are frequent, and impact the quantity and quality of sleep, leading to an increase in morbidity. Insomnia is generally defined as being a "sleep insatisfaction", and can be treated pharmacologically or non pharmacologically. Considering the side effects of the pharmacological approach, as well as the possible decrease over time of the latter's efficacy, elderly patients should initially receive a non pharmacological treatment (sleep hygiene, cognitive-behavioral therapy for insomnia) for several months before initiating a pharmacological treatment including benzodiazepines (BZP) (triazolam, estazolam, temazepam, flurazepam and quazepam), non-BZP hypnotics (zaleplon, zolpidem and eszopiclone), the recently approved suvorexant (an orexine receptor antagonist), and/or melatonin receptor agonists as well as anti depressors (doxepine).

   1.3. Sleep particularities in critical care patients Patients admitted in critical care units can be extremely vulnerable to circadian rhythm disturbances, because of the gravity of their underlying diseases, as well as environmental factors such as noise and frequent therapeutic/diagnostic interventions.

   Several factors could contribute to the sleep disturbances in these patients, mainly noise, interactions with them, mechanical ventilation, pain, drugs, artificial light, fatigue, stress delirium, altered physiology, as well as their severe disease.

   Several physiological profiles are also altered, such as arterial blood pressure, pulse, temperature, spontaneous motor activity, melatonin and cortisol levels. These sleep alterations are major sources of anxiety and stress during the ICU stay.

   Sleep studies in ICU patients have found:
   * frequent arousals;
   * sleep fragmentation;
   * alteration in the circadian rhythm;
   * a majority of NREM sleep stage 2 (N2);
   * a reduction in sleep efficiency;
   * a prolonged sleep latency;
   * an absence or decrease in the NREM sleep stage 3 (N3);
   * an absence or decrease in REM sleep Melatonin secretion is also altered in sedated patients as well as mechanically ventilated patients, as reported by certain studies. In severe sepsis patients, alterations in the urinary excretion of 6-sulfatoxymelatonin (a melatonin metabolite) are noted, suggesting a role of sepsis, as well as concomitant drugs, in the pathogenesis of melatonin secretion.

   1.4. Melatonin Administration of melatonin affects sleep architecture and thermoregulation in humans, with a causal relationship existing between melatonin and somnolence, which could be induced by thermoregulation mechanisms. This confirms the hypothesis that the initiation of melatonin secretion could contribute to the increase of somnolence as well as the increase in sleep that happens as the evening goes on.

   The diurnal administration of exogenous melatonin (when it is absent endogenously) induces sleep in humans. The levels of endogenous melatonin decrease with age, which could lead certain elderly patients to complain of bad sleep quality.

   Human studies have shown that the exogenous administration of melatonin stimulates the induction and maintenance of sleep. The increase of neuronal activity in the SCN is secondary to an increase in the endogenous nocturnal melatonin secretion. The synthesis and secretion of melatonin are parallel to the sleep rhythm, and are necessary to regulate the sleep/wake cycle by inhibiting the part of the brain responsable for the wakefulness function of the hypothalamus.

   Various melatoninergic agonists are now available to treat sleep disorders:
   * Ramelteon, for the treatment of insomnia due to difficult initiation of sleep;
   * Agomelatin, for the treatment of depression and its associated sleep disorders;
   * Tasimelteon, which seems to be effective for the treatment of the transitory insomnia due to jet lag The potential of melatonin as a hypnotic and chronobiotic agent makes its agonists good candidates for the induction of physiological sleep (in cases of insomnia and circadian rhythm alterations). They could also treat comorbid insomnia while having positive effects on a wide range of neurological, psychiatric, metabolic and cardiovascular disorders.

   Melatonin is perhaps one of the best approaches to sleep disorders, since it treats not only wake/sleep disorders, but also regulates the physiological rhythms, allowing for a better synchronized internal clock. It could be considered as a "soft and natural" treatment since it mimics the effects of a molecule which is already present in the human body.

   1.5. Pharmacogenetic of chronodisruption and its pharmacological treatment A certain number of well studied genes seem to be important to initiate and maintain the circadian rhythm, such as the CLOCK gene (Circadian Locomotor Output Cycles Kaput) which codes for proteins affecting the persistence and length of a circadian cycle; BMAL1 (Brain and Muscle AryL hydrocarbon receptor nuclear translocator-like) which is a transcription factor; PER1, PER2 and PER3 which are negative elements in the circadian transcription cycle, interacting with other regulator proteins by transporting them into the nucleus; CRY1 and CRY2 (CRYptochromes) which are also negative elements that inhibit the CLOCK-mediated transcription; and the orphan nuclear receptor RevErbA which plays an important role in the regulation of CLOCK and BMAL1's expression. The variations in the expression of all these genes can lead to variations in physiological functions and sleep architecture.

   1.6. Conclusion To this day, a small number of studies have evaluated the effect of melatonin on the modifications of the characteristics of sleep in critical care units, with mostly a small studied population. However, no study has been realized on a large population, nor has it evaluated the association between genetic factors and response to treatment, hence the originality of our study.
2. Study Objectives

Primary objectives:

* Modifications of the sleep characteristics in critical care patients
* Incidence of delirium
* Degree of agitation in patients

Secondary objectives: evaluate the effect of gene polymorphism on:

* sleep characteristics
* response to melatonin
* critical care complications
* cognitive function when waking up/at critical care discharge
* respiratory function
* endocrine function
* cardiac function
* body temperature

ELIGIBILITY:
Inclusion Criteria:

* Patients or their parents who have signed an informed consent allowing us to exploit and analyse their clinical, biological and pharmacological data (see Appendix 1)
* Patients staying more than 48 hours in ICU (acute ICU confusion occurs in the 48-72h following admission)
* Drugs affecting sleep architecture (co-variables):

  * Opiates: increase N2, decrease REM
  * NSAIDs: reduce sleep efficacy, increase arousal
  * Beta blockers: insomnia, REM sleep disappearance
  * Corticosteroids (varies according to half life and dose): REM sleep disappearance, induce awakening, stimulant effect
  * Haloperidol: increases sleep efficacy, increases N2 duration
* Respiratory assistance: ventilated patients v/s non ventilated patients (co-variables)
* Patients presenting with delirium or sleep disorders at admission will not be excluded, but a note will be taken on the baseline case report form (CRF)

Exclusion Criteria:

* Patients less than 18 years old
* Patients with central neurological disease: post traumatic patients, Parkinson disease, patients presenting with CVA, patients with neurodegenerative diseases, etc.
* Patients taking drugs capable of altering or inducing delirium:

  * Atypical antipsychotics (olanzapine, risperidone, etc.), which increase sleep efficacy, total sleep time, and NREM sleep, and reduce prevalence of ICU psychosis
  * BZD-like drugs (zolpidem, zopiclone) which induce delirium
* Melatonin allergy
* Any disorders capable of altering oral melatonin absorption (e.g. intestinal occlusion)
* Predicted ICU stay of less than 24 hours (e.g. post surgical monitoring)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2018-11-15 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Total sleep time | 14 days or ICU discharge, whichever came first
  total time spent sleeping in ICU (in minutes)

SECONDARY OUTCOMES:
REM sleep latency | 14 days or ICU discharge, whichever came first
  time from onset of sleep to REM sleep (in minutes) using an actigraph
Fragmentation index | 14 days or ICU discharge, whichever came first
  Determine how fragmented an ICU patient's sleep is using an actigraph
Sleep efficacy | 14 days or ICU discharge, whichever came first
  ratio of the total time spent asleep (total sleep time) in a night compared to the total amount of time spent in bed (minutes) using an actigraph
Incidence of delirium in ICU | 14 days or ICU discharge, whichever came first
  Evaluate delirium in ICU using the CAM-ICU (confusion assessment method for the ICU) scale (presence or absence of delirium)
Degree of agitation of patients | 14 days or ICU discharge, whichever came first
  Evaluate agitation using the RASS (Richmond Agitation Sedation Scale) scale using a total score ranging from -5 to +4, the lower being a more sedated patient and the higher a more agitated patient
Gene polymorphism | 14 days or ICU discharge, whichever came first
  Evaluate the effect of gene polymorphism (CLOCK gene, BMAL) using a genetic test, on sleep characteristics, response to melatonin and critical care complications
Sleep latency | 14 days or ICU discharge, whichever came first
  time from trying to sleep to actually falling asleep (in minutes)

CONTACTS AND LOCATIONS:
Locations (1):
- Hotel Dieu de France, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Knauert MP, Malik V, Kamdar BB. Sleep and sleep disordered breathing in hospitalized patients. Semin Respir Crit Care Med. 2014 Oct;35(5):582-92. doi: 10.1055/s-0034-1390080. Epub 2014 Oct 29. PMID 25353103
- [Background] Gandhi AV, Mosser EA, Oikonomou G, Prober DA. Melatonin is required for the circadian regulation of sleep. Neuron. 2015 Mar 18;85(6):1193-9. doi: 10.1016/j.neuron.2015.02.016. Epub 2015 Mar 5. PMID 25754820
- [Background] Gabor JY, Cooper AB, Crombach SA, Lee B, Kadikar N, Bettger HE, Hanly PJ. Contribution of the intensive care unit environment to sleep disruption in mechanically ventilated patients and healthy subjects. Am J Respir Crit Care Med. 2003 Mar 1;167(5):708-15. doi: 10.1164/rccm.2201090. PMID 12598213
- [Background] Pisani MA, Friese RS, Gehlbach BK, Schwab RJ, Weinhouse GL, Jones SF. Sleep in the intensive care unit. Am J Respir Crit Care Med. 2015 Apr 1;191(7):731-8. doi: 10.1164/rccm.201411-2099CI. PMID 25594808
- [Background] Jones CR, Huang AL, Ptacek LJ, Fu YH. Genetic basis of human circadian rhythm disorders. Exp Neurol. 2013 May;243:28-33. doi: 10.1016/j.expneurol.2012.07.012. Epub 2012 Jul 28. PMID 22849821
- [Background] Ely EW, Inouye SK, Bernard GR, Gordon S, Francis J, May L, Truman B, Speroff T, Gautam S, Margolin R, Hart RP, Dittus R. Delirium in mechanically ventilated patients: validity and reliability of the confusion assessment method for the intensive care unit (CAM-ICU). JAMA. 2001 Dec 5;286(21):2703-10. doi: 10.1001/jama.286.21.2703. PMID 11730446
- [Background] Huang H, Jiang L, Shen L, Zhang G, Zhu B, Cheng J, Xi X. Impact of oral melatonin on critically ill adult patients with ICU sleep deprivation: study protocol for a randomized controlled trial. Trials. 2014 Aug 18;15:327. doi: 10.1186/1745-6215-15-327. PMID 25135124